CLINICAL TRIAL: NCT05144282
Title: The Analysis of Association of Retinopathy of Prematurity, Gut Microbiome Profile, and Systemic Inflammation
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201902088A3
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Retinopathy of Prematurity; Microbiome
Keywords: Retinopathy of prematurity; microbiome; very low birth weight; inflammatory cytokine
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Stool samples will be collected within 1-week-of-age and then every 2 weeks (± 3 days) until PMA 40 weeks or until infant is discharged from our hospital. Samples are collected from diapers and immediately stored briefly at 4°C, and frozen at -80°C until analyzed. The microbiome profiling will be processed either by 16S rRNA sequencingor shotgun metagenomic sequencing.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- premature baby without ROP (Group 1): ROP: retinopathy of prematurity
- ROP without treatment (Group 2): ROP: retinopathy of prematurity
- ROP with anti-VEGF treatment (Group 3): ROP: retinopathy of prematurity
  Interventions: Procedure: intravitreal injection of anti VEGF
- ROP with laser photocoagulation treatment (Group 4): ROP: retinopathy of prematurity
  Interventions: Procedure: laser photocoagulation

INTERVENTIONS:
Procedure: intravitreal injection of anti VEGF — The treatment for ROP was either primary intravitreal injection (IVI) of anti-vascular endothelial growth factor (anti-VEGF).
  Groups: ROP with anti-VEGF treatment (Group 3)
Procedure: laser photocoagulation — The treatment for ROP was either primary laser photocoagulation.
  Groups: ROP with laser photocoagulation treatment (Group 4)

SUMMARY:
Study Aims

1. Understanding the gut microbiome profile in very low birth weight infants with or without ROP. The onset and aggravation of ROP and their relationship with gut microbiome will be examined.
2. Understanding the serum inflammatory cytokine profile in these infants and its relationship with the onset and progression of ROP. Their changes and association with the other systemic disorders such as NEC or RDS or sepsis will be explored.
3. Examiningthe associations amongmicrobiome profile and serum inflammatory cytokines and their relationship with ROP clinical features (prematurity without ROP, ROP without treatment, and ROP with treatment) in the study participant

DETAILED DESCRIPTION:
Background In recent decades, severeretinopathy of prematurity (ROP) and the proportion of ROP needing treatment is increasing. These conditions are due to the fact that more premature infants now could surviveowing to the improvement in neonatology. Since ROP isa leading cause of blindness in children, how to deal with these severely affected eyes becomes a major challenge.

In recent years, growing evidence support that exposure to infection and inflammation increases risk of ROP and these exposures are considered key contributors to the pathogenesis of ROP. These exposures, which are modifiable, have gained interest among researchers.

The microbiome are symbiotic organisms living inside human bodies. They are most abundant in human gastrointestinal tracts and play a fundamental role in host inflammatory and immunity physiology. The gut microbiome is most extensively studied, and reports showed that they play a role not only in gastrointestinal inflammatory diseases, but also in extra-gastrointestinal conditions.

Recent data have shown that microbiome changes may involve in the pathogenesisof ophthalmic diseasessuch as uveitis, but its role in ROP has not been explored. Since ROP is closely related to inflammation, and that the gut microbiome has a significant role in the modulation of both systemic and ocular inflammatory pathways, we are interested to know whether there is association between ROP, microbiome, and systemic inflammation. Whether the microbiome profile is different in ROP and no-ROP neonates is worth exploring. Also, it is important to see whether the onset of ROP is related to the systemic inflammation status. To the best of our knowledge, there are no report on such topic, therefore our current study is designed to answer this question.

Methods Very low birth weight preterm infantsborn in our hospital from August 2020to July 2023 will be enrolled into study. Infants who has major or congenital GI anomaly will be excluded. ROP screening protocol and categorization will follow the international standards. DNA will be extracted from the stool samples and underwent microbiome profiling either by 16S rRNA or shotgun metagenomic sequencing. Blood samples from the routine blood examinations will beanalyzed by an immunoassay to reveal the level of systemic inflammation (IL-1 alpha/beta, IL-10, IL-13 and so on). Statistical analysis will be performed and the associations among ROP features, gut microbiome, and serum inflammatory cytokines will be explored.

Study Aims

1. Understanding the gut microbiome profile in very low birth weight infants with or without ROP. The onset and aggravation of ROP and their relationship with gut microbiome will be examined.
2. Understanding the serum inflammatory cytokine profile in these infants and its relationship with the onset and progression of ROP. Their changes and association with the other systemic disorders such as NEC or RDS or sepsis will be explored.
3. Examiningthe associations amongmicrobiome profile and serum inflammatory cytokines and their relationship with ROP clinical features (prematurity without ROP, ROP without treatment, and ROP with treatment) in the study participant

ELIGIBILITY:
Inclusion Criteria:

* All GA<37 weeks preterm infants with birth weight (BW) between 500 and 1500 grams born in Linkou of Chung Gung Memorial Hospital from August 2020 to July 2023 will be enrolled into study after obtaining informed consent from their parent within 1-week-of-age.

Exclusion Criteria:

* Preterm infants who has major or congenital gastrointestional (GI) anomaly (eg. trisomy 13, trisomy 18, esophageal or intestinal atresia, GI obstruction, meconium peritonitis with prenatal bowel perforation, etc.).

Ages: 1 Day to 1 Week | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All GA<37 weeks preterm infants with birth weight (BW) between 500 and 1500 grams born in Linkou of Chung Gung Memorial Hospital from August 2020 to July 2023 will be enrolled into study after obtaining informed consent from their parent within 1-week-of-age.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2020-08-15 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Gut Microbiome | 2020-2023
  Understanding the gut microbiome profile in very low birth weight infants with or without ROP. The onset and aggravation of ROP and their relationship with gut microbiome will be examined.
Serum Inflammatory Cytokine | 2020-2023
  Understanding the serum inflammatory cytokine profile in these high-risk infants and its relationship with the onset and progression of ROP. Their changes and association with the other systemic disorders such as NEC or RDS or sepsis will be explored.
Microbiome Profile And Serum Inflammatory Cytokines And Their Relationship with ROP | 2020-2023
  Examining the associations among microbiome profile and serum inflammatory cytokines and their relationship with ROP clinical features in the study participants (patients with prematurity without ROP, patients with ROP without treatment, and patients with ROP and treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Wu WeiChi, M.D., PhD., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Department of Ophthalmology, Chang Gung Memorial Hospital., Taoyuan District, Linkou, Taiwan